CLINICAL TRIAL: NCT00151619
Title: Regional and Systemic Hemodynamic Effects of a Long-term Administration of Amlodipine in Patients With Chronic Heart Failure Treated With a Combination of Enalapril, Furosemide and Digoxin
Brief Title: Effects of Amlodipine in the Management of Chronic Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFSSAPS 960723; LOC-H/95-02; CIC0203/005
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Chronic Heart Failure
Keywords: Calcium channel blockers; Heart failure; Hemodynamics
MeSH Terms: conditions — Heart Failure | interventions — Amlodipine

INTERVENTIONS:
Drug: Amlodipine

SUMMARY:
Patients with congestive heart failure are usually treated with a combination of an ACE inhibitor (or an AT1 blocking agent), a diuretic and a beta-blocker. However, some patients remain symptomatic despite an optimal treatment with these drugs. In patients who also have coronary heart disease, nitrates or some calcium-channel blockers could help to relieve symptoms. Therefore, the aim of our study is to evaluate the additional benefit induced by a second generation calcium-channel blocker, amlodipine, in patients with chronic heart failure who remain symptomatic despite an optimal treatment.

DETAILED DESCRIPTION:
In patients with congestive heart failure, a treatment with ACE inhibitor combined with digoxin and a diuretic has shown benefits on morbidity and mortality. However, 40% of these patients have persistant symptoms. The rationale for the use of calcium channel blockers in patients with chronic heart failure lies in their vasodilating action, antiischemic effect, ability to reduce left ventricular diastolic dysfunction. The objective of our study is to evaluate the regional and systemic hemodynamic, hormonal and vascular effects and the tolerance to stress test of a 3-months treatment with amlodipine. Patients with stable chronic heart failure (III/IV NYHA) and treated with a combination of enalapril, furosemide and digoxin will be randomized to receive amlodipine 5 or 10 mg or a placebo for a 3-months period.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Chronic heart failure with New York Heart Association class III or IV.
* Ischemic or dilated cardiopathy known for at least 3 months
* Systolic arterial pressure > 110 mmHg under treatment
* Stroke volume between 20 and 40% under treatment
* Informed written consent

Exclusion Criteria:

* History of allergy to one of the studied pharmaceutical classes
* History of troubles in ventricular rythm (tachycardia, fibrillation) or acute heart failure
* Chronic renal, hepatic or respiratory failure
* Diabetes
* Valvulopathy
* Myocarditis,constrictive pericarditis
* Life prognosis < 6 months due to a non cardiac pathology
* Absence of woman contraception, pregnancy, breast-feeding
* Treatment with calcium channel blockers or antiarrythmics class IC
* Unstable patient under standardized treatment
* Unable to do a stress test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 1999-02-10 (Actual); Primary Completion 2001-09-06 (Actual)

PRIMARY OUTCOMES:
Humeral blood flow

SECONDARY OUTCOMES:
Systemic hemodynamics:
- Systolic and diastolic arterial pressures
- Heart rate and cardiac output
- Systolic and diastolic left ventricular diameters
- Ambulatory measure of arterial pressure
- Isovolumic relaxation time, pulmonary venous flow
Regional hemodynamics:
- Carotid, humeral and femoral arterial diameters and flows
- Arterial compliance
- Renal and hepatosplanchnic blood flow
Stress test
Biological variables: ionogram, hormonal and cytokines plasma concentrations
Functional well-being measure on a Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bellissant, MD, PhD, Principal Investigator — CHU Rennes
Locations (2):
- France (2):
  - Service de Réanimation Médicale - Hôpital Raymond Poincaré, Garches
  - Service de Réadaptation Cardio-Vasculaire - Clinique St Yves, Rennes

REFERENCES:
- [Background] Elkayam U, Shotan A, Mehra A, Ostrzega E. Calcium channel blockers in heart failure. J Am Coll Cardiol. 1993 Oct;22(4 Suppl A):139A-144A. doi: 10.1016/0735-1097(93)90478-j. PMID 8376684
- [Background] Cohn JN, Johnson G, Ziesche S, Cobb F, Francis G, Tristani F, Smith R, Dunkman WB, Loeb H, Wong M, et al. A comparison of enalapril with hydralazine-isosorbide dinitrate in the treatment of chronic congestive heart failure. N Engl J Med. 1991 Aug 1;325(5):303-10. doi: 10.1056/NEJM199108013250502. PMID 2057035
- [Background] Packer M, O'Connor CM, Ghali JK, Pressler ML, Carson PE, Belkin RN, Miller AB, Neuberg GW, Frid D, Wertheimer JH, Cropp AB, DeMets DL. Effect of amlodipine on morbidity and mortality in severe chronic heart failure. Prospective Randomized Amlodipine Survival Evaluation Study Group. N Engl J Med. 1996 Oct 10;335(15):1107-14. doi: 10.1056/NEJM199610103351504. PMID 8813041